CLINICAL TRIAL: NCT05686811
Title: Comparative Effect of Myofascial Release Therapy and Post Isometric Relaxation Technique on Pain and Functional Disability in Patients With Tension Type Headache
Brief Title: Tension Type Headache, Myofascial Release Therapy , Post Isometric Relaxation Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-UOL-/226-09/2022
Record Dates: First submitted 2022-10-24; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Neck Pain
Keywords: Myofascial release therapy
MeSH Terms: conditions — Neck Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: To compare the effects of myofascial release therapy and post isometric relaxation technique on pain and functional disability in patients with tension type headache
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial release therapy (Active Comparator): This group will receive routine physical therapy with myofascial release therapy.This protocol will be given for 3 alternative days per week. Each session will be of 40 minutes. Data will be calculated at baseline , at 2nd and at 4th week.
  Interventions: Other: Myofascial release therapy therapy
- post isometric relaxation technique (Experimental): This group will receive routine physical therapy with post isometric relaxation technique.This protocol will be given for 3 alternative days per week. Each session will be of 40 minutes. Data will be calculated at baseline , at 2nd and at 4th week.
  Interventions: Other: Post isometric relaxation technique

INTERVENTIONS:
Other: Myofascial release therapy therapy — Group A was treated with myofascial release therapy and routine physical therapy. For routine physical therapy subjects will first applied TENS, hot pack and neck isometric exercises then myofascial release therapy will be given. For myofascial release therapy subjects was in the supine or possibly sitting position, the examiner was seated at the head of the table, the examiner was used his right thumb to palpate (using flat palpation) the upper trapezius muscles from medial to lateral to establish if any MTrPs are present. The entire mass of the upper trapezius muscle is lifted by the supraspinatus muscle and grasped with a pincer grasp. The muscles at this point rotate between the thumb and forefinger to detect the delicate location of the trigger point. Treatment session longs for 10 minutes of myofascial release on each side
  Arms: Myofascial release therapy
Other: Post isometric relaxation technique — This group will receive routine physical therapy with myofascial release therapy.This protocol will be given for 3 alternative days per week. Each session will be of 40 minutes. Data will be calculated at baseline , at 2nd and at 4th week.
  Arms: post isometric relaxation technique

SUMMARY:
COMPARATIVE EFFECTS OF MYOFASCIAL RELEASE THERAPY AND POST ISOMETRIC RELAXATION TECHNIQUE ON PAIN AND FUNCTIONAL DISABILITY IN PATIENTS WITH TENSION-TYPE HEADACHE

DETAILED DESCRIPTION:
Tension-type headache (TTH) is the most common type of primary headache, typically presenting as a bilateral, non-throbbing headache with mild to moderate intensity. Patients with tension-type headache often report band-like tightness and increased tenderness of the pericranial muscles. Use of myofascial release technique and post isometric relaxation technique is believed to reduce the pain and improve the functional disability.

ELIGIBILITY:
Inclusion Criteria:

* • Age range 25-45years14

  * Both male and females
  * Suffer from tension type headache more than three months
  * Head pain on bilateral location
  * may suffer from photophobia, phonophobia
  * Pericranial tiredness
  * not getting enough exercise or sleep

Exclusion Criteria:

* • History of teeth clenching or grinding

  * Cardiovascular disease
  * Pregnancy
  * arthritis in the neck
  * being overweight

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Numerical pain rating scale | at the end of 4th week
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Mateen, MS(msk), Principal Investigator — University of Lahore
Locations (1):
- Abdul Mateen, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No